CLINICAL TRIAL: NCT02467660
Title: Meditation or Health & Wellness Education Via Internet for Adults 50-80 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Barry S. Oken, MD, PhD, Oregon Health and Science University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 11847
Record Dates: First submitted 2015-05-20; First posted 2015-06-10 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Stress, Physiological; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness; Health

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Online Mindfulness Meditation Training (Experimental): Weekly 1-hr online training and daily meditation for 30-45 min for 6 wks
  Interventions: Behavioral: Mindfulness Meditation
- Online Health & Wellness Education (Experimental): 6-week training entails completing weekly 1-hour online training and listening to educational podcasts for 30-45 minutes per day
  Interventions: Behavioral: Health & Wellness Education
- Wait List Control (No Intervention): No training

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Using study-provided iPod device to listen to guided meditations daily
  Arms: Online Mindfulness Meditation Training
Behavioral: Health & Wellness Education — Using study-provided iPod device to listen to educational podcasts daily
  Arms: Online Health & Wellness Education

SUMMARY:
1. Telephone Eligibility Screening
2. Baseline Visit, includes online questionnaires, physical measures, cognitive tasks, voice recordings, physical recordings of brain waves, heart rate, breathing rate, and sweat during computer tasks. Collect saliva samples, questionnaire data, and respond to handheld device that rings randomly for the seven days following the visit.
3. Randomized to receive (a) an internet-based Mindfulness Meditation program, (b) an internet-based Health & Wellness Education program, or (c) no training. IF assigned to receive a training program, participants complete weekly one-hour online trainings and daily home practice for 6 weeks
4. Endpoint Visit (same as Baseline), scheduled 8 weeks after Baseline
5. All participants receive Meditation and Education programs after the Endpoint Visit
6. Online questionnaire follow-up 6 months after the Endpoint

DETAILED DESCRIPTION:
The primary aim of this research project is to evaluate whether an internet-based mindfulness meditation training improves cognition and resilience in stressed older adults. Dr. Oken specializes in evaluating the effects of stress on the human body, and he plans to use advanced statistical analyses to create a "multi-domain physiologic measure." This means study staff will collect biological data, including electroencephalogram (EEG, brainwaves), blood pressure, heart rate, breathing rate, and saliva samples. The investigator hypothesizes that when he statistically combines all of these together, he will have a measure that correlates with self-rated (survey) measures of resilience and stress.

Participants will undergo a telephone screening to determine eligibility, and then they will fill out online questionnaires before their Baseline Visit at the lab. Study staff will take physical measurements (i.e. height, weight, vision), administer short cognitive tasks that measure attention and memory, and collect biological data (listed above) during several different tasks. Some of the tasks are very simple, such as breath counting and listening to an audio recording of a podcast. And some of the tasks are intended to be more stressful, such as one that presents difficult math problems. The investigator hopes to induce stress so that study staff can measure resilience by evaluating how long it takes participants to return to a biological baseline, such as their usual blood pressure. In total, the visit is approximately 3 ½ hours long.

After the Baseline, participants are sent home with a handheld device that administers random 5-minute assessments, as well as tubes to collect saliva, for the seven days following the in-lab visit. Participants will also fill out short questionnaires about daily events over these seven days. Once data collection is complete, participants will come into the lab to return the device and samples and learn whether they have been randomized to receive the internet-based mindfulness meditation training (40% chance), an internet-based health & wellness education program (40% chance), or a non-active waitlist (20% chance). All participants will be informed before the study begins that they will have access to the meditation and education materials once their participation is complete. Participants receiving the meditation and education will complete a one-hour online training each week for six weeks, and they will use an iPod to listen to guided meditations or educational podcasts (depending on group assignment) for 30-45 minutes per day. The iPod tracks their home practice, and they will return it at the end of the study. All participants will receive a weekly call from study staff to check in about whether they have experienced any health changes and, if applicable, how the meditation or education program is going.

Eight weeks after the Baseline Visit, participants will again fill out online questionnaires and come back to the lab for an Endpoint Visit, which is very similar to the Baseline. They will again collect saliva samples and complete assessments on a handheld device for two days following the visit. They will mail the samples and device back to the lab and then receive access to both internet-based training programs and associated audio recordings. Participants will then be asked to fill out online questionnaires one last time 6 months after the Endpoint Visit.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50 and 80 years old
* Be stable on all medications for at least 2 months and willing to NOT change medications for the duration of the study
* Have access to a computer with internet in order to complete online questionnaires three separate times and complete 1-hour trainings once per week for six weeks
* Willing to travel to OHSU for a total of three times
* Willing to follow the study protocol, including completely weekly internet-based trainings and doing 30-45 minutes of home practice daily for 6 weeks IF randomly assigned to receive the meditation or education trainings

Exclusion Criteria:

* Have any significant medical or neurological diseases, such as major organ failure, insulin-dependent diabetes, or active cancer
* Have significant untreated depression
* Have significant visual or hearing impairment
* Take certain medications in the last 2 months, such as neuroleptics or steroids
* Have prior experience with mediation classes or other mind-body classes (e.g. yoga or tai chi) within the past 2 years
* Have had a regular meditation practice in the past 30 days
* Be gone for more than one full week during study participation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Golden Stroop Cognitive Task Total Score | Change from Baseline in Stroop score at 8 weeks
  Measures selective attention, cognitive flexibility, and processing speed
Heart Rate Variability | Change from Baseline in Heart Rate Variability at 8 weeks
  Used as a measure of resiliency to determine how quickly a participant returns to baseline following an experimental stressor
Composite multi-domain physiologic measure | Change in multiple measures from Baseline at 8 weeks
  ECG, EEG, Respiration, self-report questionnaires

SECONDARY OUTCOMES:
Rey Auditory Verbal Learning Task Total Score | Change from Baseline in AVLT scores at 8 weeks
  Evaluates short-term auditory-verbal memory, rate of learning, learning strategies, retroactive and proactive interference, presence of confabulation of confusion in memory processes, retention of information, and differences between learning and retrieval
Verbal Fluency Total Score | Change from Baseline in Verbal Fluency score at 8 weeks
  Measures executive function
Letter Number Sequencing Total Score | Change from Baseline in Letter Number Sequencing score at 8 weeks
  Measures executive function
Systolic and Diastolic Blood Pressure | Change from Baseline in Systolic and Diastolic Blood Pressure at 8 weeks
  Used as a measure of resiliency to determine how quickly a participant returns to baseline following an experimental stressor
Respiration Rate | Change from Baseline in Respiration Rate at 8 weeks
  Used as a measure of resiliency to determine how quickly a participant returns to baseline following an experimental stressor
Salivary Cortisol Levels | Change from Baseline in Cortisol Levels at 8 weeks
  Measures general stress from baseline to endpoint and it's also used as a measure of resiliency to determine how quickly a participant returns to baseline following an experimental stressor; Several samples are taken during Baseline and Endpoint Assessments (8 weeks apart), and four samples are collected each day for two days following the Baseline and two days following the Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Oken, MD, MS, Principal Investigator — Oregon Health and Science University
Locations (1):
- Hatfield Research Center, Portland, Oregon, United States